CLINICAL TRIAL: NCT07184398
Title: Use of a Cysteine-rich Whey Protein Isolate (Immunocal®) in Post COVID-19 Cognitive Impairment
Brief Title: Use of a Cysteine-rich Whey Protein Isolate in Post COVID-19 Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Libre seccional Cali (Other)
Collaborators: Immunotec Inc. (Industry)
Responsible Party: Principal Investigator, Ingrid Mena, Neuropsychologist, Universidad Libre seccional Cali
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 860013798-5
Record Dates: First submitted 2025-09-09; First posted 2025-09-19 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: COVID-19 (SARS-CoV-2 Infection)
Keywords: covid-19; oxidative stress; brain fog; cognitive disorder; cysteine; whey protein
MeSH Terms: conditions — COVID-19; Mental Fatigue; Cognitive Dysfunction | interventions — Methods

STUDY DESIGN:
Intervention Model Description: This open-label study evaluates the use of a cysteine-rich whey protein isolate (Immunocal®) in patients with post-COVID-19 cognitive impairment. Oxidative stress and glutathione depletion are believed to contribute to persistent neurological and respiratory symptoms. Since direct glutathione supplementation is poorly absorbed, Immunocal® provides bioavailable cystine, which is converted to cysteine-the rate-limiting precursor for intracellular glutathione synthesis. Daily supplementation aims to restore redox balance, reduce neuroinflammation, and improve cognitive performance, fatigue, and quality of life in COVID-19 survivors. Outcomes include validated cognitive tests, fatigue scales, and biomarkers of oxidative stress and inflammation to explore clinical and mechanistic effects.
Who Masked: Participant
Masking Description: This is an open-label study. No masking will be applied. All participants, care providers, and investigators will be aware of the treatment being administered. Outcome assessors will also be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- No intervention (No Intervention): Participants will receive no specific nutritional supplementation or rehabilitation beyond routine medical follow-up. This group serves as the natural history comparator for cognitive outcomes.
- Neuropsychological rehabilitation (Active Comparator): Participants will undergo a structured neuropsychological rehabilitation program targeting memory, attention, and executive function deficits associated with post-COVID-19 cognitive impairment. Standardized cognitive exercises and behavioral strategies will be applied over the intervention period.
  Interventions: Behavioral: Cognitive rehabilitation workshops
- Immunocal® (Cysteine-Rich Whey Protein Isolate) (Experimental): CRWPI Immunocal® (Immunotec™) was administered at a dose of 20 grams (2 sachets once daily) for 12 consecutive weeks. The research team delivered Immunocal directly to the subjects and instructed them on how to mix and self-administer it.
  Interventions: Other: Intervention with Consolidated Cysteine (Immunocal) 20 g per day

INTERVENTIONS:
Other: Intervention with Consolidated Cysteine (Immunocal) 20 g per day — CRWPI Immunocal® (Immunotec™) was administered at a dose of 20 grams (2 sachets once daily) for 12 consecutive weeks. The research team delivered Immunocal directly to the subjects and instructed them on how to mix and self-administer it.
  Arms: Immunocal® (Cysteine-Rich Whey Protein Isolate)
Behavioral: Cognitive rehabilitation workshops — Neuropsychological rehabilitation consisted of in-person group sessions for 40 adults (18 years or older) to work on cognitive functions such as memory and attention. Each session lasted 45 minutes. These sessions were held three times a week for a period of 12 weeks.
  Arms: Neuropsychological rehabilitation

SUMMARY:
Abstract Background: Post-COVID-19 cognitive impairment (PCCI), characterized by deficits in attention, memory, and executive functioning, remains a major challenge among patients with long COVID. Oxidative stress is a key contributor to this condition. Cysteine-rich whey protein isolate (CRWPI), such as Immunocal®, enhances intracellular glutathione production and may offer neuroprotective benefits.

Objective: To evaluate the efficacy of Immunocal® supplementation on cognitive function, particularly attention and memory, and functional performance in individuals with ICCP.

Methods: A randomized, controlled, parallel-group trial was conducted in Cali, Colombia, with 120 adults recovering from COVID-19 with mild to moderate cognitive impairment. Participants were randomly assigned to three groups: (1) immune® supplementation (CRWPI) (20 g/day), (2) neuropsychological rehabilitation, or (3) no intervention (control), for 12 weeks. Cognitive outcomes were assessed using the Montreal Cognitive Assessment (MoCA) and the NEUROPSI attention and memory test. Physical endurance was measured using the 30-second foot test (STST). Clinical symptoms evaluated through a medical assessment form, before and after the intervention, were also taken into account. Results: Both the Immunocal® and neurorehabilitation groups showed statistically significant improvements in all attention subdomains and memory types compared to the control. Immunocal® produced greater gains in divided attention and working memory, suggesting a specific advantage in cognitive domains sensitive to oxidative stress. STST performance was also significantly improved in the Immunocal® group. No significant improvements were seen in the control group.

Conclusion: Immunocal® supplementation significantly improves cognitive performance, comparable to structured neurorehabilitation, in individuals with ICCP. It also shows potential to improve physical endurance, clinical symptoms, and reduce fatigue. These findings support the integration of Immunocal® as a non-pharmacological intervention for cognitive dysfunction related to long COVID.

DETAILED DESCRIPTION:
Study Design and Participants This randomized, controlled, parallel-group trial included subjects at least 18 years of age in Cali, Colombia, who recovered from COVID-19 infection and presented with mild to moderate cognitive impairment and no history of Immunocal administration. Subjects with a history of cerebrovascular or cardiovascular disease and current or previous use of Immunocal were excluded from screening. Ethical approval was obtained from the IRB of the Universidad Libre and informed consent was obtained.

Sampling and protocol A consecutive non-probabilistic sampling was performed. For this study, a target sample of 120 subjects was selected to achieve a 95% confidence level. A double-blind randomization process was used to divide subjects into three groups of 40 participants as follows: 1. CRWPI (Immunocal®) supplementation; 2. Structured neuropsychological rehabilitation (Neurorehabilitation), and no intervention (control).

A group of neuropsychologists with experience in the application of cognitive tools and neuropsychological rehabilitation were responsible for the evaluation and management of the neuropsychological phase of the study. Neuropsychological rehabilitation consisted of 45-minute face-to-face group sessions that were conducted three times a week over a 12-week period. After 12 weeks, a neuropsychological evaluation was completed on each subject.

CRWPI Immunocal® (Immunotec ™) was administered at a dose of 20 grams (2 sachets once daily) for 12 consecutive weeks. The research team delivered the Immunocal directly to the subjects and instructed them how to mix and self-administer it.

Pre-test cognitive functioning was assessed using NEUROPSI attention and memory, while only NEUROPSI attention and memory were used to assess the same cognitive domains at 12 weeks.

The main objective of NEUROPSI Attention and Memory is to assess a broad spectrum of cognitive functions, including spatial, temporal and personal orientation; attention and concentration; working memory; verbal and visual memory, and executive and motor functions. The NEUROPSI Attention and Memory test considers age and schooling for the acquisition of quantitative and qualitative data and classifies amnesic and attentional alterations into four different categories.

The 30-second sit-stand (STST) test is a widely used assessment designed to assess lower-body strength and functional endurance.19 It measures how many complete stops a person can complete from a seated position in 30 seconds, without using their arms for support. This test provides valuable information about muscle strength and balance, making it a practical tool for monitoring physical performance and the effectiveness of interventions such as exercise programs or nutritional supplements. STST is often used to assess fatigue in the muscles of the lower extremities and trunk. This test was performed on all available participants after the intervention period was completed.

The participants were also evaluated before and after the intervention by the doctors of the research group, through a medical assessment form where all clinical symptoms due to the virus were recorded.

ELIGIBILITY:
Inclusion:

* Adults ≥18 years with confirmed prior COVID-19
* with persistent cognitive symptoms
* able to complete testing
* and willing to consent.

Exclusion:

* Pre-existing dementia or major psychiatric illness
* whey protein allergy - participation in another cognitive trial
* severe hepatic/renal/metabolic disease, pregnancy
* or any condition interfering with participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Change in Cognitive Function | 12 weeks
  Cognitive performance will be assessed using a standardized neuropsychological test battery evaluating memory, attention, and executive function. Scores will be compared from baseline to the end of the intervention period.

SECONDARY OUTCOMES:
Change in Functional Capacity (Sit-to-Stand Test) | 12 weeks
  Functional capacity will be measured by the 30-second sit-to-stand test. The number of repetitions completed will be compared between baseline and study completion.

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Mena, Neuropsychologist, Principal Investigator — Universidad Libre
Locations (1):
- Doctor's office, Cali, Valle del Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-09-16): https://cdn.clinicaltrials.gov/large-docs/98/NCT07184398/Prot_SAP_ICF_003.pdf